CLINICAL TRIAL: NCT02994134
Title: Exercise, Cognitive Function and Neuroplasticity in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joyce Rios Gomes Osman, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20161059
Record Dates: First submitted 2016-12-01; First posted 2016-12-15 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate intensity exercise. (Active Comparator): Moderate intensity aerobic exercise intervention (delivered at 55-64% age-predicted maximal heart rate), 4 times per week for 4 weeks.
  Interventions: Behavioral: Moderate intensity exercise.
- High intensity exercise (Experimental): High intensity aerobic exercise intervention (delivered at 65%-90% age-predicted maximal heart rate), 4 times per week for 4 weeks.
  Interventions: Behavioral: High intensity exercise.

INTERVENTIONS:
Behavioral: Moderate intensity exercise. — Moderate intensity aerobic exercise intervention (delivered at 55-64% age-predicted maximal heart rate), 4 times per week for 4 weeks.
  Arms: Moderate intensity exercise.
Behavioral: High intensity exercise. — High intensity aerobic exercise intervention (delivered at 65-90% age-predicted maximal heart rate), 4 times per week for 4 weeks.
  Arms: High intensity exercise

SUMMARY:
The overall goal of the proposed study is to compare the effects of 4 weeks of moderate or high intensity aerobic exercise on neuroplasticity, cognitive performance and gait and postural control in sedentary healthy adults.

DETAILED DESCRIPTION:
The primary aim of the study is to compare the effects of a moderate intensity aerobic exercise intervention (delivered at 55-64% age-predicted maximal heart rate) with a high intensity aerobic exercise intervention (delivered at 65%-90% age-predicted maximal heart rate) on measures that probe cortical synaptic plasticity using transcranial magnetic stimulation (TMS) in sedentary healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged 18-70 years old
* Primary language is English
* Sedentary (defined as not engaging in purposeful physical activity more than 2 times over the last two months)
* Exercise clearance

Exclusion Criteria:

* Presence of cognitive, neurologic or orthopedic conditions that could affect performance of the testing and training procedures
* History of migraines.
* History of fainting spells of unknown or undetermined etiology that might constitute seizures
* History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform) EEG or family history of treatment resistant epilepsy
* Any current history of a psychiatric illness
* Any unstable medical condition
* No medication is an absolute exclusion from TMS. Medications will be reviewed by the Principal Investigator and a decision about inclusion will be made based on the following:

  * The subject's past medical history, drug dose, history of recent medication changes or duration of treatment, and combination with other CNS active drugs.
  * The published TMS guidelines review medications to be considered with TMS (Rossi, Hallett, Rossini, Pascual-Leone, & Safety of TMS Consensus Group, 2009).
* Any metal in the brain, skull or elsewhere unless approved by the responsible MD
* Any medical devices (i.e. Cardiac pacemaker, deep brain stimulator, medication infusion pump, cochlear implant, vagal nerve stimulator)
* Intracranial lesion
* Substance abuse or dependence within the past six months Subjects who, in the Investigator's opinion, might not be suitable for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Change in cortical synaptic plasticity using transcranial magnetic stimulation (TMS) from baseline to post-exercise. | Baseline, 4 weeks
  Plasticity with TMS

CONTACTS AND LOCATIONS:
Overall Officials: Joyce R Gomes Osman, PT, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No